CLINICAL TRIAL: NCT00109642
Title: Investigating the Role of Norepinephrine in Emotional Processing Through Alpha-2 Adrenergic Receptor Modulation
Brief Title: The Role of Norepinephrine in Emotional Processing
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050147; 05-M-0147
Record Dates: First submitted 2005-04-29; First posted 2005-05-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-08

CONDITIONS: Psychopathy; Mental Disorders
Keywords: Amygdala; Orbitofrontal Cortex; Yohimbine; Emotion; Guanfacine; Norepinephrine; Healthy Volunteer
MeSH Terms: conditions — Antisocial Personality Disorder; Mental Disorders

SUMMARY:
This study will examine the role of a brain chemical called norepinephrine in thinking, decision-making, and emotional processing. After norepinephrine is released from a brain cell, it binds to another brain cell's receptor. Some of the receptors it binds to are called alpha-2 adrenergic receptors. This study will use medicines called yohimbine and guanfacine to look at the function of norepinephrine in the brain when it binds to the alpha-2 adrenergic receptors. Yohimbine increases norepinephrine's function and guanfacine decreases its function.

Healthy volunteers between 20 and 50 years of age who do not have heart disease, high blood pressure, psychiatric illness, or other serious medical conditions and who are not allergic to lactose may be eligible for this study. Candidates are screened with a medical and psychiatric history, physical examination, neuropsychological testing, blood and urine tests and electrocardiogram. Women are screened with a urine pregnancy test.

Participants are given a pill of yohimbine, guanfacine, or placebo and undergo the following tests and procedures:

* Blood pressure and heart rate measurements: Blood pressure and heart rate are measured before the medication is taken and several times after.
* Blood draws: Blood is drawn before the medicine is taken and 90 minutes after to measure levels of norepinephrine and the hormone cortisol.
* Neurocognitive testing: Participants do neurocognitive tasks on the computer for up to 90 minutes. The tasks involve looking at pictures or words on a screen and responding according to instructions given.
* Magnetic resonance imaging (MRI): Patients may undergo neurocognitive testing MRIs. This test uses a strong magnetic field and radio waves to show changes in brain activity. The subject lies on a table that slides into a narrow cylinder (the MRI scanner). Images of the brain are obtained while the subject performs the computer tasks.

DETAILED DESCRIPTION:
An understanding of the role of specific neurotransmitters in the neurocognitive functions mediating emotional processing is essential for the understanding and treatment of mood and anxiety disorders. One such disorder, currently regarded as untreatable, is psychopathy. Psychopathy has been linked with noradrenergic and amygdala disturbances. However, an understanding of the functional significance of the noradrenergic system in humans remains in its infancy. The goal of this protocol is to use targeted noradrenergic manipulations (yohimbine and guanfacine) in conjunction with specific neurocognitive and neuroimaging paradigms to consider the role of norepinephrine in reward and punishment processing. In particular, we wish to evaluate the hypothesis that increased norepinephrine levels following the administration of yohimbine will lead to enhanced formation and processing of stimulus-reward and stimulus-punishment associations, while decreased norepinephrine levels following the administration of guanfacine will reduce the formation and processing of stimulus-reward and stimulus-punishment associations. In addition, we aim to examine the hypothesis that increased norepinephrine levels will lead to increased neural response in the amygdala during either the formation, or processing, of stimulus-reinforcement associations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Participants will be males and females, 20-50 years of age.

IQ: IQ, as measured by 4 subscales from the Wechsler Adult Intelligence Scale-Revised (WAIS-R), must be greater than 80.

Medication status: No current use of any psychotropic medication or benzodiazepine.

EXCLUSION CRITERIA:

Because factors such as psychiatric disease, or CNS disease, can influence functional brain activity, these factors are exclusionary:

* Psychiatric History: Participants will be assessed using DSM-IV criteria via standardized psychiatric interviews conducted by trained examiners (SCID). All participants will be free of any current or past major affective disorder, psychotic disorder, substance dependence, anorexia, somatoform disorder, or anxiety disorders with the exception of specific phobias.
* Severe acute and chronic medical illnesses (e.g. cardiac disease, diabetes, epilepsy).
* CNS disease: Known history of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), other central nervous system disease, or history of head trauma which resulted in a persistent neurologic deficit or loss of consciousness greater than 3 minutes.
* Currently on regular medication that would interfere with study results. This includes alpha and beta adrenergic medications, other anti-hypertensive medications, glucocorticoid and mineralocorticoid medications, and medications causing sedation or stimulation. For example, current use of tylenol or ibuprofen is permitted, while current use of benadryl or methylphenidate is not. Use of oral contraceptive pills is permitted.
* Currently breast feeding or pregnant (as documented by pregnancy testing at screening or at days of the challenge studies).

Additional exclusion criteria for fMRI studies:

* Metal or electronic objects: Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.
* Claustrophobia: participants will be questioned about potential discomfort in being in an enclosed space, such as an MRI scanner.
* Body weight - to reduce the likelihood of significant orthostasis from guanfacine, participants must weigh 60kg or greater. Those weighing less than 60 kg will be excluded.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216
Dates: Start 2005-04-26; Primary Completion 2009-03-15 (Actual); Study Completion 2009-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R. Neural systems for recognizing emotion. Curr Opin Neurobiol. 2002 Apr;12(2):169-77. doi: 10.1016/s0959-4388(02)00301-x. PMID 12015233
- [Background] Arnsten AF. Adrenergic targets for the treatment of cognitive deficits in schizophrenia. Psychopharmacology (Berl). 2004 Jun;174(1):25-31. doi: 10.1007/s00213-003-1724-3. Epub 2003 Dec 19. PMID 15205875
- [Background] Aron AR, Fletcher PC, Bullmore ET, Sahakian BJ, Robbins TW. Stop-signal inhibition disrupted by damage to right inferior frontal gyrus in humans. Nat Neurosci. 2003 Feb;6(2):115-6. doi: 10.1038/nn1003. No abstract available. PMID 12536210